CLINICAL TRIAL: NCT06878781
Title: Standardized Meals With Different Macronutrient Ratios on the Postprandial Metabolome and Metabolic Flexibility
Brief Title: Postprandial Metabolome and Metabolic Flexibility
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Medicina Genomica (Other Government)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Principal Investigator, Berenice Palacios-Gonzalez, PhD, Instituto Nacional de Medicina Genomica
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 467
Record Dates: First submitted 2024-04-08; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Fasting; Postprandial Hyperglycemia; Lipid Metabolism Disorders; Glucose Metabolism Disorders; Insulin Sensitivity
Keywords: metabolic flexibility; postprandial response; mixed meals
MeSH Terms: conditions — Fasting; Hyperglycemia; Lipid Metabolism Disorders; Glucose Metabolism Disorders; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Enrolled subjects are followed every week for one month. At each visit, a questionnaire assesses daily time-activity patterns. Dietary intake is assessed by a food frequency questionnaire and a multi-step 24-hour dietary recall. Subjects will then be randomized to receive the metabolic challenges in a different order. The procedures will be performed before (fasting; 8-10 hours) and after (postprandial) consumption of the metabolic challenges. Capillary blood samples are obtained in the morning after an 8-hour fasting and after test meal consumption. Once the drop of blood is formed, it is placed directly into the CardioCheck Plus® cassette to determine glucose triglyceride, LDL-cholesterol, HDL-cholesterol, and total cholesterol. A second drop of capillary blood shall be placed on a filter paper. Indirect fasting calorimetry is also performed. After the indirect calorimetry, the metabolic and hormonal response to the test meal is performed.
Who Masked: Investigator
Masking Description: There will be a single-blind principal investigator (PI). All results will be coded and will remain closed until the study is completed. The PI will remain blind to the results until the codes are opened at the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- High carbohydrate challenge (Experimental): High carbohydrate challenge should be consumed within 15 minutes. After 5 minutes of rest, indirect calorimetry will be postprandially, lasting 30 minutes.
  Capillary blood shall be obtained at the following times: 15-30-45-60-90 and 120 min after ingestion of food.
  Interventions: Other: High carbohydrate challenge
- High lipid challenge (Experimental): High lipid challenge should be consumed within 15 minutes. After 5 minutes of rest, indirect calorimetry will be postprandially, lasting 30 minutes. Capillary blood shall be obtained at the following times: 15-30-45-60-90 and 120 min after ingestion of food.
  Interventions: Other: High lipid challenge
- High protein challenge (Experimental): High protein challenge should be consumed within 15 minutes. After 5 minutes of rest, indirect calorimetry will be postprandially, lasting 30 minutes. Capillary blood shall be obtained at the following times: 15-30-45-60-90 and 120 min after ingestion of food.
  Interventions: Other: High proteinchallenge

INTERVENTIONS:
Other: High carbohydrate challenge — Capillary blood samples will be obtained in the morning after an overnight 8-hour fasting; then, an indirect fasting calorimetry will be performed. After the indirect calorimetry, the metabolic and hormonal response to the test meal is performed. The nutritional composition of the standardized meal is shown below. Energy, 479.6 kcal; Carbohydrate, 83.6%; Lipids, 12.4%, and Protein, 4.0% (70 g of hot cake, 100 g of mango, 270 ml of peach nectar, and 40 g of strawberry jam). The food challenge should be consumed within 15 minutes. After 5 minutes of rest, indirect calorimetry will be postprandially, lasting 30 minutes. Capillary blood shall be obtained at the following times: 15-30-45-60-90 and 120 min after ingestion of food.
  Arms: High carbohydrate challenge
Other: High lipid challenge — Capillary blood samples will be obtained in the morning after an overnight 8-hour fasting; then, an indirect fasting calorimetry will be performed. After the indirect calorimetry, the metabolic and hormonal response to the test meal is performed. The nutritional composition of the standardized meal is shown below. Energy, 1043.4 kcal; Carbohydrate, 4.9%; Lipids, 86.8%, and Protein, 8.3% (60 g of manchego cheese, 25 g of egg, white, dried, 24 g of bacon, 5 ml of oil, 65 g of cream cheese, 70 g of cream, and 16 g of poblano pepper). The food challenge should be consumed within 15 minutes. After 5 minutes of rest, indirect calorimetry will be postprandially, lasting 30 minutes. Capillary blood shall be obtained at the following times: 15-30-45-60-90 and 120 min after ingestion of food.
  Arms: High lipid challenge
Other: High proteinchallenge — Capillary blood samples will be obtained in the morning after an overnight 8-hour fasting; then, an indirect fasting calorimetry will be performed. After the indirect calorimetry, the metabolic and hormonal response to the test meal is performed. The nutritional composition of the standardized meal is shown below. Energy, 441.3 kcal; Carbohydrate, 1.6%; Lipids, 5.1%, and Protein, 93.3% (2 scoop Isopure Zero Carb, 180 g of chicken breast, 20 g of lettuce and 24 g of ham turkey breast). The food challenge should be consumed within 15 minutes. After 5 minutes of rest, indirect calorimetry will be postprandially, lasting 30 minutes. Capillary blood shall be obtained at the following times: 15-30-45-60-90 and 120 min after ingestion of food.
  Arms: High protein challenge

SUMMARY:
Metabolic flexibility is a process in which the body can switch energy substrates in different physiological states. This flexibility plays an important role in an individual's health because losing it increases the risk of obesity, metabolic syndrome, insulin resistance, and type 2 diabetes. Considering that humans spend most of their awakening hours in a postprandial (PP) state, an organism's metabolic flexibility (MF) to respond to a standardized meal's consumption would provide information on the individual's metabolic health. The PP response to glucose following an oral glucose tolerance test or consumption of a high-carbohydrate meal is well described; however, few studies assess the FM and PP metabolome using mixed meals with different macronutrients. The investigators address how metabolic flexibility and metabolome change after consuming standardized meals with different macronutrient ratios. Data collection includes clinical and diet information, indirect calorimetry, and capillary blood sampling during fasting and after consumption of standardized meals. Samples are collected weekly for one month. The data will determine the metabolic flexibility and metabolome after consuming standardized meals with different macronutrient ratios.

DETAILED DESCRIPTION:
Enrolled subjects are followed every week for one month. At each visit, a questionnaire assesses daily time activity patterns relevant to energy expenditure, general health status, including infectious symptoms, and confirmation of basic social and demographic characteristics. Dietary intake is assessed by a food frequency questionnaire and a multi-step 24-hour dietary recall for quantitative analysis. If symptoms of infection are present, participants are treated with ad-hoc broad antibiotics. Anthropometrics are obtained. Subjects will then be randomized to receive the metabolic challenges in a different order. The procedures will be performed before (fasting; 8-10 hours) and after (postprandial) consumption of the metabolic challenges. Capillary blood samples (40µ) are obtained in the morning after an 8-hour fasting and after test meal consumption. To obtain the capillary blood sample, sterilize the ring finger with alcohol and allow it to dry. Then, puncture the area with a sterile 2 mm long lancet. Once the drop of blood is formed, it is placed directly into the CardioCheck Plus® cassette to determine glucose triglyceride, LDL-cholesterol, HDL-cholesterol, and total cholesterol. A second drop of capillary blood shall be placed on a filter paper (S&S 903) until a circle of filter paper is filled with blood to saturate the paper throughout its thickness. Insulin concentration shall be determined following the protocol for dried blood, which is standardized in the laboratory. Indirect fasting calorimetry is also performed. After the indirect calorimetry, the metabolic and hormonal response to the test meal is performed.

Each challenge should be consumed within 15 minutes. After 5 minutes of rest, indirect calorimetry will be postprandially, lasting 30 minutes. Capillary blood shall be obtained at the following times: 15-30-45-60-90 and 120 min after ingestion of food.

Nutrient composition of standardized meal and meal example.

* High carbohydrate challenge: Energy, 479.6 kcal; Carbohydrate, 83.6%; Lipids, 12.4% and Protein, 4.0% (70 g of hot-Cake, 100 g of mango, 270 ml of peach nectar, and 40 g of strawberry jam)
* High lipid challenge: Energy, 1043.4 kcal; Carbohydrate, 4.9%; Lipids, 86.8%, and Protein, 8.3% (60 g of manchego cheese, 25 g of egg, white, dried, 24 g of bacon, 5 ml of oil, 65 g of cream cheese, 70 g of cream, and 16 g of poblano pepper)
* High protein challenge: Energy, 441.3 kcal; Carbohydrate, 1.6%; Lipids, 5.1%, and Protein, 93.3% (2 scoop Isopure Zero Carb, 180 g of chicken breast, 20 g of lettuce and 24 g of ham turkey breast)

Determination of metabolites in dried blood To determine the concentration of metabolites (amino acids and acyl-carnitines), a circle of 3 mm diameter shall be punched out of the filter paper and placed in a 96-well plate. Add 100 µl of the acyl-carnitine and amino acid standards from the NeoBase PerkinElmer kit. Subsequently, follow the manufacturer's instructions for determining metabolites by liquid chromatography coupled to mass spectrometry (LC-MS).

Determination of the respiratory quotient (RQ) To determine the respiratory quotient (RQ= VmaxCO2/ VmaxO2) and lipid and carbohydrate oxidation examinations, the Cardio Coach CO2 Vmax Encore 29 System calorimeter software (Korr, Inc, UT, USA) will be used according to the instructions of the supplier. Examinations are invariably performed in the morning (8:00-9:00 am) in a thermoneutral environment with controlled pressure, humidity, and temperature, with the patient supine but awake. The investigators examine a maximum of two subjects per day. Oxygen consumption and carbon dioxide production were obtained using a canopy and were monitored continuously for 30 minutes. The initial 10 minutes of the measurement are discarded for the calculation to ensure greater data homogeneity. O2 consumption and CO2 production will be recorded continuously for 30 min. VO2 and VCO2 values will be used in the equation proposed by Weir (Energy Expenditure = [3.941(VO2) + 1.11(VCO2)] x 1440 min/day), considered as the standard method [34]. Additionally, one day before the test, subjects are instructed to fast for 8 hours and not engage in physical activity or consume caffeine the day before the exam. All participants will be asked to eat the same dinner the night before each test. Dinner provides 15% of the daily energy intake; 20 g of protein, 7 g of lipids, and 34 g of carbohydrates)

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years of age and under 30 years of age;
* without active drug addictions: smoking, alcoholism, and/or drug addiction;
* in female subjects: regular menstrual cycles;
* give written consent for their inclusion in the study.

Exclusion Criteria:

* subjects with any pathology that requires medication or special treatment, such as type 2 diabetes mellitus, high blood pressure, dyslipidemia, polycystic ovary syn-drome, autoimmune, thyroid, kidney, neurological diseases, and cancer;
* pregnant or lactating women;
* subjects with problems with chewing, salivation, and swallowing.

Elimination criteria:

* subjects who only have samples (blood and calorimetry) from one study period (fasting or postprandial);
* subjects who only have samples (blood and calorimetry) of a metabolic challenge;
* subjects who have an infection at the scheduled appointment;
* subjects who withdraw their informed consent

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-18 (Estimated)

PRIMARY OUTCOMES:
Metabolic Flexibility Assessed by Respiratory Quotient (RQ) and Substrate Oxidation | Once a week for three weeks
  Metabolic flexibility will be assessed by measuring the respiratory quotient (RQ) and substrate oxidation during fasting and postprandial states. RQ values are expected to range from 0.70 to 0.80 during fasting and vary during the postprandial period depending on the food consumed: 0.87-1.00 for the high-carbohydrate challenge, 0.70-80 for the high-fat challenge, and 0.81-0.90 for the high-protein challenge. Measurements will be conducted using the Cardio Coach CO2 Vmax Encore 29 System Calorimeter. Oxygen consumption (VO2) and carbon dioxide production (VCO2) values will be used to calculate energy expenditure using Weir's equation: Energy Expenditure = [3.941(VO2) + 1.11(VCO2)] × 1440 min/day.

SECONDARY OUTCOMES:
Postprandial Glucose Levels | Once a week for three weeks
  Measure of postprandial glucose concentration (ml/dL) after meal intake.
Postprandial Triglyceride Levels | Once a week for three weeks
  Measure of postprandial triglyceride concentration (mg/dL) after meal intake.
Postprandial Acyl Carnitines Levels | Once a week for three weeks
  Measure of postprandial acyl carnitines concentration (µmol/L) after meal intake.
Postprandial Amino Acid Levels | Once a week for three weeks
  Measure of postprandial amino acid concentration (µmol/L) after meal intake.

CONTACTS AND LOCATIONS:
Overall Officials: Berenice Palacios-Gonzalez, PhD, Principal Investigator — National Institute of Genomic Medicine; Noemi Meraz-Cruz, PhD, Principal Investigator — Universidad Nacional Autonoma de Mexico
Locations (1):
- Berenice Palacios-Gonzalez, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schonknecht YB, Crommen S, Stoffel-Wagner B, Coenen M, Fimmers R, Holst JJ, Simon MC, Stehle P, Egert S. Acute Effects of Three Different Meal Patterns on Postprandial Metabolism in Older Individuals with a Risk Phenotype for Cardiometabolic Diseases: A Randomized Controlled Crossover Trial. Mol Nutr Food Res. 2020 May;64(9):e1901035. doi: 10.1002/mnfr.201901035. Epub 2020 Apr 15. PMID 32223057
- [Background] Weinisch P, Fiamoncini J, Schranner D, Raffler J, Skurk T, Rist MJ, Romisch-Margl W, Prehn C, Adamski J, Hauner H, Daniel H, Suhre K, Kastenmuller G. Dynamic patterns of postprandial metabolic responses to three dietary challenges. Front Nutr. 2022 Sep 22;9:933526. doi: 10.3389/fnut.2022.933526. eCollection 2022. PMID 36211489
- [Background] Kelley DE, Mandarino LJ. Fuel selection in human skeletal muscle in insulin resistance: a reexamination. Diabetes. 2000 May;49(5):677-83. doi: 10.2337/diabetes.49.5.677. PMID 10905472
- [Background] Delgadillo-Velazquez JA, Nambo-Venegas R, Patino N, Meraz-Cruz N, Razo-Azamar M, Guevara-Cruz M, Fonseca M, Pale Montero LE, Ibarra-Gonzalez I, Vela-Amieva M, Vadillo-Ortega F, Palacios-Gonzalez B. Metabolic flexibility during normal pregnancy allows appropriate adaptation during gestation independently of BMI. Clin Nutr ESPEN. 2021 Aug;44:254-262. doi: 10.1016/j.clnesp.2021.06.007. Epub 2021 Jun 19. PMID 34330475
- [Background] Gupta RD, Ramachandran R, Venkatesan P, Anoop S, Joseph M, Thomas N. Indirect Calorimetry: From Bench to Bedside. Indian J Endocrinol Metab. 2017 Jul-Aug;21(4):594-599. doi: 10.4103/ijem.IJEM_484_16. PMID 28670546
- [Background] Lepine G, Tremblay-Franco M, Bouder S, Dimina L, Fouillet H, Mariotti F, Polakof S. Investigating the Postprandial Metabolome after Challenge Tests to Assess Metabolic Flexibility and Dysregulations Associated with Cardiometabolic Diseases. Nutrients. 2022 Jan 21;14(3):472. doi: 10.3390/nu14030472. PMID 35276829
- [Background] Muoio DM. Metabolic inflexibility: when mitochondrial indecision leads to metabolic gridlock. Cell. 2014 Dec 4;159(6):1253-62. doi: 10.1016/j.cell.2014.11.034. PMID 25480291
- [Background] Zeevi D, Korem T, Zmora N, Israeli D, Rothschild D, Weinberger A, Ben-Yacov O, Lador D, Avnit-Sagi T, Lotan-Pompan M, Suez J, Mahdi JA, Matot E, Malka G, Kosower N, Rein M, Zilberman-Schapira G, Dohnalova L, Pevsner-Fischer M, Bikovsky R, Halpern Z, Elinav E, Segal E. Personalized Nutrition by Prediction of Glycemic Responses. Cell. 2015 Nov 19;163(5):1079-1094. doi: 10.1016/j.cell.2015.11.001. PMID 26590418
- [Background] Bansal S, Buring JE, Rifai N, Mora S, Sacks FM, Ridker PM. Fasting compared with nonfasting triglycerides and risk of cardiovascular events in women. JAMA. 2007 Jul 18;298(3):309-16. doi: 10.1001/jama.298.3.309. PMID 17635891
- [Background] Nishida T, Tsuji S, Tsujii M, Arimitsu S, Haruna Y, Imano E, Suzuki M, Kanda T, Kawano S, Hiramatsu N, Hayashi N, Hori M. Oral glucose tolerance test predicts prognosis of patients with liver cirrhosis. Am J Gastroenterol. 2006 Jan;101(1):70-5. doi: 10.1111/j.1572-0241.2005.00307.x. PMID 16405536
- [Background] Vis, D.J., et al., Analyzing metabolomics-based challenge tests. Metabolomics, 2015. 11(1): p. 50-63.
- [Background] Krug S, Kastenmuller G, Stuckler F, Rist MJ, Skurk T, Sailer M, Raffler J, Romisch-Margl W, Adamski J, Prehn C, Frank T, Engel KH, Hofmann T, Luy B, Zimmermann R, Moritz F, Schmitt-Kopplin P, Krumsiek J, Kremer W, Huber F, Oeh U, Theis FJ, Szymczak W, Hauner H, Suhre K, Daniel H. The dynamic range of the human metabolome revealed by challenges. FASEB J. 2012 Jun;26(6):2607-19. doi: 10.1096/fj.11-198093. Epub 2012 Mar 16. PMID 22426117
- [Background] LaBarre JL, Singer K, Burant CF. Advantages of Studying the Metabolome in Response to Mixed-Macronutrient Challenges and Suggestions for Future Research Designs. J Nutr. 2021 Oct 1;151(10):2868-2881. doi: 10.1093/jn/nxab223. PMID 34255076
- [Background] Yu EA, Yu T, Jones DP, Ramirez-Zea M, Stein AD. Metabolomic Profiling After a Meal Shows Greater Changes and Lower Metabolic Flexibility in Cardiometabolic Diseases. J Endocr Soc. 2020 Aug 25;4(11):bvaa127. doi: 10.1210/jendso/bvaa127. eCollection 2020 Nov 1. PMID 33134764
- [Background] Sebedio, j.-l. and S. Polakof, Using metabolomics to identify biomarkers for metabolic diseases: Analytical methods and applications. 2015. p. 145-166.
- [Background] Adamska-Patruno E, Samczuk P, Ciborowski M, Godzien J, Pietrowska K, Bauer W, Gorska M, Barbas C, Kretowski A. Metabolomics Reveal Altered Postprandial Lipid Metabolism After a High-Carbohydrate Meal in Men at High Genetic Risk of Diabetes. J Nutr. 2019 Jun 1;149(6):915-922. doi: 10.1093/jn/nxz024. PMID 31049566
- [Background] van den Broek TJ, Bakker GCM, Rubingh CM, Bijlsma S, Stroeve JHM, van Ommen B, van Erk MJ, Wopereis S. Ranges of phenotypic flexibility in healthy subjects. Genes Nutr. 2017 Dec 6;12:32. doi: 10.1186/s12263-017-0589-8. eCollection 2017. PMID 29225708
- [Background] Fiamoncini J, Rundle M, Gibbons H, Thomas EL, Geillinger-Kastle K, Bunzel D, Trezzi JP, Kiselova-Kaneva Y, Wopereis S, Wahrheit J, Kulling SE, Hiller K, Sonntag D, Ivanova D, van Ommen B, Frost G, Brennan L, Bell J, Daniel H. Plasma metabolome analysis identifies distinct human metabotypes in the postprandial state with different susceptibility to weight loss-mediated metabolic improvements. FASEB J. 2018 Oct;32(10):5447-5458. doi: 10.1096/fj.201800330R. Epub 2018 May 2. PMID 29718708
- [Background] Kardinaal AF, van Erk MJ, Dutman AE, Stroeve JH, van de Steeg E, Bijlsma S, Kooistra T, van Ommen B, Wopereis S. Quantifying phenotypic flexibility as the response to a high-fat challenge test in different states of metabolic health. FASEB J. 2015 Nov;29(11):4600-13. doi: 10.1096/fj.14-269852. Epub 2015 Jul 21. PMID 26198450
- [Background] Yu EA, Yu T, Jones DP, Martorell R, Ramirez-Zea M, Stein AD. Macronutrient, Energy, and Bile Acid Metabolism Pathways Altered Following a Physiological Meal Challenge, Relative to Fasting, among Guatemalan Adults. J Nutr. 2020 Aug 1;150(8):2031-2040. doi: 10.1093/jn/nxaa169. PMID 32597983
- [Background] Shrestha A, Mullner E, Poutanen K, Mykkanen H, Moazzami AA. Metabolic changes in serum metabolome in response to a meal. Eur J Nutr. 2017 Mar;56(2):671-681. doi: 10.1007/s00394-015-1111-y. Epub 2015 Dec 10. PMID 26658764
- [Background] Moriya T, Satomi Y, Kobayashi H. Metabolomics of postprandial plasma alterations: a comprehensive Japanese study. J Biochem. 2018 Feb 1;163(2):113-121. doi: 10.1093/jb/mvx066. PMID 29040577
- [Background] Mathew S, Krug S, Skurk T, Halama A, Stank A, Artati A, Prehn C, Malek JA, Kastenmuller G, Romisch-Margl W, Adamski J, Hauner H, Suhre K. Metabolomics of Ramadan fasting: an opportunity for the controlled study of physiological responses to food intake. J Transl Med. 2014 Jun 6;12:161. doi: 10.1186/1479-5876-12-161. PMID 24906381
- [Background] Yu EA, Le NA, Stein AD. Measuring Postprandial Metabolic Flexibility to Assess Metabolic Health and Disease. J Nutr. 2021 Nov 2;151(11):3284-3291. doi: 10.1093/jn/nxab263. PMID 34293154
- [Background] Bastarrachea RA, Laviada-Molina HA, Nava-Gonzalez EJ, Leal-Berumen I, Escudero-Lourdes C, Escalante-Araiza F, Peschard VG, Veloz-Garza RA, Haack K, Martinez-Hernandez A, Barajas-Olmos FM, Molina-Segui F, Buenfil-Rello FA, Gonzalez-Ramirez L, Janssen-Aguilar R, Lopez-Munoz R, Perez-Cetina F, Gaytan-Saucedo JF, Vaquera Z, Cornejo-Barrera J, Castillo-Pineda JC, Murillo-Ramirez A, Diaz-Tena SP, Figueroa-Nunez B, Gonzalez-Lopez L, Salinas-Osornio RA, Valencia-Rendon ME, Angeles-Chimal J, Santa-Olalla Tapia J, Remes-Troche JM, Valdovinos-Chavez SB, Huerta-Avila EE, Han X, Orozco L, Rodriguez-Ayala E, Weintraub S, Gallegos-Cabrales EC, Cole SA, Kent JW Jr. Deep Multi-OMICs and Multi-Tissue Characterization in a Pre- and Postprandial State in Human Volunteers: The GEMM Family Study Research Design. Genes (Basel). 2018 Nov 2;9(11):532. doi: 10.3390/genes9110532. PMID 30400254
- [Background] Wopereis S, Stroeve JHM, Stafleu A, Bakker GCM, Burggraaf J, van Erk MJ, Pellis L, Boessen R, Kardinaal AAF, van Ommen B. Multi-parameter comparison of a standardized mixed meal tolerance test in healthy and type 2 diabetic subjects: the PhenFlex challenge. Genes Nutr. 2017 Aug 29;12:21. doi: 10.1186/s12263-017-0570-6. eCollection 2017. PMID 28861127
- [Background] Smith RL, Soeters MR, Wust RCI, Houtkooper RH. Metabolic Flexibility as an Adaptation to Energy Resources and Requirements in Health and Disease. Endocr Rev. 2018 Aug 1;39(4):489-517. doi: 10.1210/er.2017-00211. PMID 29697773
- [Background] Patricio, B.P., et al., Normal menstrual cycle. Intech Open, 2019. doi:10.5772/intechopen. 79876
- [Background] Ibarra-Gonzalez I, Rodriguez-Valentin R, Lazcano-Ponce E, Vela-Amieva M. Metabolic screening and metabolomics analysis in the Intellectual Developmental Disorders Mexico Study. Salud Publica Mex. 2017 Jul-Aug;59(4):423-428. doi: 10.21149/8668. PMID 29211263
- [Background] Mtaweh H, Tuira L, Floh AA, Parshuram CS. Indirect Calorimetry: History, Technology, and Application. Front Pediatr. 2018 Sep 19;6:257. doi: 10.3389/fped.2018.00257. eCollection 2018. PMID 30283765
- [Background] Goodpaster BH, Sparks LM. Metabolic Flexibility in Health and Disease. Cell Metab. 2017 May 2;25(5):1027-1036. doi: 10.1016/j.cmet.2017.04.015. PMID 28467922
- [Background] Morris C, O'Grada CM, Ryan MF, Gibney MJ, Roche HM, Gibney ER, Brennan L. Modulation of the lipidomic profile due to a lipid challenge and fitness level: a postprandial study. Lipids Health Dis. 2015 Jul 1;14:65. doi: 10.1186/s12944-015-0062-x. PMID 26123789